CLINICAL TRIAL: NCT07270718
Title: The Influence of Beetroot Powder at a Dose of 20 g on Blood Pressure, Microcirculation, and Biochemical Markers in Men With Arterial Hypertension.SVEKLA2025.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Collaborators: Saratov State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-07/24
Record Dates: First submitted 2025-11-26; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-09

CONDITIONS: Hypertensive Heart Disease Without (Congestive) Heart Failure
Keywords: exogenous nitrate, nitric oxide, blood pressure, endothelial dysfunction, beetroot
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plus SVEKLA (Experimental): Powder SVEKLA 20 g (800 mg NOx)
  Interventions: Dietary Supplement: Plus SVEKLA
- No SVEKLA (No Intervention)

INTERVENTIONS:
Dietary Supplement: Plus SVEKLA — The first time in the Russian Federation beetroot powder (20 g equivalent 800 mg NOx) in clinical trial in patients with hypotension disease
  Arms: Plus SVEKLA

SUMMARY:
Objective: to evaluate the effectiveness of using a food product, dry finely dispersed beetroot powder in a dose of 20 g, containing 800 mg of nitrate (NO3-), in relation to the regulation of blood pressure in men with hypertension who reached the target blood pressure level while taking optimal antihypertensive therapy.

Characteristics of the study: randomized, open, and cross-sectional. Relevance of the study Currently, it is recognized that vasodilatory endothelial dysfunction due to impaired synthesis and bioavailability of endogenous nitric oxide (NO) is a characteristic change in patients with arterial hypertension (AH) and plays one of the key roles in the development and progression of this pathology.

Nitrate (NO3-), contained in food products, the highest content of which is found in beetroot, is converted into NO in the body after consumption, which can have a positive effect on the state of the cardiovascular system and lead to a decrease in blood pressure. Indeed, this assumption has been confirmed in various clinical studies. The results of the conducted studies demonstrate the positive effect of beetroot juice enriched with NO3- on the functional parameters of the cardiovascular system, in particular, the level of SAD and DBP, vasodilator function, endothelium and arterial stiffness, both in patients with hypertension and conditionally healthy people.

However, most of the studies conducted in this field either include a relatively small number of subjects with hypertension, or do not have a cross-sectional design, which is a limitation in formulating unambiguous conclusions about the positive effect of taking beetroot enriched with NO3- on lowering blood pressure in this category of patients. Moreover, the effect of beetroot juice on the functional state of the peripheral arterial bed (terminal muscular arteries, distributive and precapillary arterioles) remains unexplored, which, due to the increased bioavailability of NO by the vascular wall, may be expressed in a decrease in arterial stiffness, a decrease in smooth muscle cell tone (MMC) and a decrease in total peripheral vascular resistance, which will have a positive effect on tissue homeostasis. It is relevant to study the effect of course intake of beetroot enriched with NO3- on the functional state of all arterial links and regulation of blood pressure in patients with hypertension.

Research materials and methods The study will be performed on the basis of the Laboratory of Microcirculation and Regional Blood Circulation of the Department of Fundamental and Applied Aspects of Obesity and the Center for Coordination of Fundamental Scientific Activities of the Federal State Budgetary Institution "NMIC TPM" of the Ministry of Health of the Russian Federation. The study is planned to include 60 men aged 18-60 years with hypertension who reached the target blood pressure level according to office measurement and daily blood pressure monitoring (SMAD) on the background of regular intake of AGT.

Research design The study will consist of two screening stages and one main stage (Figure 1). Patients will be divided into 2 equal groups of 30 men using simple randomization using the closed envelope method. The first group will be assigned a one-week course of daily intake of dry fine beetroot powder in a dose of 20 g containing 800 mg of NO3- (food product), the second group will continue regular intake of AGT. After 7 days, the crossing will be performed: patients of the first group will continue to receive regular AGT, and patients of the second group will receive a food product. At each stage, all participants undergo blood pressure and heart rate (HR) measurements, anthropometry, basic research methods* and SMAD. The total duration of the study will be 14-16 days.

ELIGIBILITY:
Inclusion Criteria:

* A history of hypertension with achievement of the target blood pressure level according to the SMAD while taking regular AGT;
* signing informed consent to participate in the study.

Exclusion Criteria:

* coronary heart disease, including angina pectoris and myocardial infarction; cerebrovascular disease, including acute cerebrovascular accident and transient ischemic attack; obliterating atherosclerosis of peripheral vessels, revascularization in any vascular basin; cardiomyopathy; secondary forms of hypertension; type 1 or 2 diabetes mellitus, impaired glucose tolerance; inflammatory bowel diseases; organ transplantation; oncological, mental illnesses; diffuse connective tissue diseases in the anamnesis;
* BMI ≥30 kg/m2;
* symptoms of heart failure;
* acute infectious diseases at the time of inclusion in the study and within 1 month prior to inclusion in the study;
* Exacerbation of chronic non-communicable diseases;
* alcoholism, taking narcotic drugs;
* allergic and undesirable reactions to foods containing beetroot and egg white in the anamnesis;
* refusal to continue participating in the study

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — men
Enrollment: 60 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Blood pressure decrease | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- National Medical Research Center for Preventive Medicine, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No